CLINICAL TRIAL: NCT03762772
Title: A Phase I Study to Assess Safety, Pharmacokinetics, and Pharmacodynamics of a Vaginal Insert Containing Tenofovir Alafenamide and Elvitegravir
Brief Title: Safety, PK, and PD Study of a Vaginal Insert Containing TAF and EVG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: Eastern Virginia Medical School (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A18-146
Record Dates: First submitted 2018-11-16; First posted 2018-12-04 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Hiv; HSV
Keywords: HIV; TAF; EVG; Prevention; Vaginal Insert
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: All participants will use a single combination TAF/EVG vaginal insert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAF/EVG vaginal insert (Experimental): Post-dose sampling at 4 and 48 hours or at 24 and 72 hours, per randomization
  Interventions: Drug: TAF/EVG Vaginal Insert

INTERVENTIONS:
Drug: TAF/EVG Vaginal Insert — 1 combination vaginal insert (20mg TAF/16mg EVG)

SUMMARY:
The purpose of this Phase I study is to assess the safety, pharmacokinetics, and pharmacodynamics of a combination vaginal insert containing tenofovir alafenamide (TAF) and elvitegravir (EVG).

This study will be the first-in-human study for a vaginally administered TAF/EVG insert and will evaluate safety, PK and PD after a single dose. It is hypothesized that the combination insert will be safe and well-tolerated by study participants and that the insert will offer an expanded window of preventive activity and a regimen with flexibility and forgiveness.

DETAILED DESCRIPTION:
This Phase I study aims to complete at least 16 healthy, non-pregnant, HIV-uninfected women aged 18-50 years who are not at risk for pregnancy and are at low risk for sexually transmitted infections (STIs) at one clinical site. The study will examine the safety, PK, PD, disintegration, and acceptability of vaginal inserts containing the combination of tenofovir alafenamide (TAF) and elvitegravir (EVG).

Participants will be randomized (1:1) into one of two sample collection time point groups:

[Timepoint group 1: 4 and 48 hours after using the single combination insert] or [Timepoint group 2: 24 and 72 hours after using the single combination insert]

There will be 5 scheduled visits:

Visit 1 (Screening/Enrollment): Volunteers will be consented and undergo tests and procedures to confirm they are eligible to continue in the study.

Visit 2 (Baseline): Once it has been confirmed that participants are eligible and willing to continue, they will be asked to complete a short baseline questionnaire about the insert. Participants will be randomized to Timepoint group 1 or Timepoint group 2 for sample collection and will then undergo baseline sampling [cervicovaginal (CV) fluid and tissue].

Visit 3 (Insert use and sampling): Participants will use a single combination insert of TAF/EVG in the clinic. Depending upon timepoint randomization, percentage disintegration of the vaginal inserts will be assessed at either 4 hours or 24 hours, and PK and PD sample collection (plasma, CV fluid, and CV tissue) will occur. Participants will also be asked to complete a short acceptability questionnaire.

Visit 4 (Post-Dose Sampling): Participants will undergo sample collection of blood for safety and PK evaluations; and CV fluid and CV tissue for PK at either 48 hours or 72 hours depending upon timepoint randomization.

Visit 5 (Post-Dose Sampling): Participants will undergo a PK sample collection (CV fluid) 7 (±2) days post dose. Participants will be asked about adverse events and concomitant medications taken. Participants will then be exited from the study, unless they have symptoms that require follow-up.

There will be 5 scheduled visits over approximately 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years, inclusive
2. General good health (by volunteer history and per investigator judgment) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, bone disease, and diabetes) and with an intact uterus and cervix.
3. History of regular menstrual cycles, by volunteer report (for cycling women)
4. History of Pap smears and follow-up consistent with standard clinical practice as outlined in the Study Manual or willing to undergo a Pap smear at Visit 1
5. Able to communicate in spoken and written English
6. Willing to give voluntary consent and sign an informed consent form
7. Willing and able to comply with protocol requirements, including abstaining from vaginal activity and product use at specified times
8. Must be protected from pregnancy by one of the following:

   * Hormonal methods, except vaginal rings and DMPA
   * Copper IUD
   * Sterilization of participant or partner
   * Consistent condom use
   * Abstinence from penile-vaginal intercourse
   * Same sex relationship
9. If in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive and has no known risk of sexually transmitted infections (STIs)

Exclusion Criteria:

1. Positive pregnancy test or plans to become pregnant during the course of the study
2. Currently breastfeeding or planning to breastfeed during the course of the study
3. History of sensitivity/allergy to any component of the study product, topical anesthetic, or to both silver nitrate and Monsel's solution
4. In the last three months, diagnosed with or treated for any STI (For HSV, ideally no outbreaks in the past year. More than two outbreaks in previous 12 month period is exclusionary.)
5. Positive test for Trichomonas vaginalis (TV), Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), HIV, or Hepatitis B surface antigen (HBsAg)
6. Symptomatic bacterial vaginosis (BV)
7. Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
8. Known blood disorder, including deep vein thrombosis (DVT) and pulmonary embolism (PE), or those that could lead to prolonged or continuous bleeding with biopsy
9. NSAIDS, systemic corticosteroids (e.g. dexamethasone), Endothelin Receptor Antagonists (e.g bosentan), antibiotics, Anticonvulsants (e.g. carbamazepine, oxcarbazepine, phenobarbital, phenytoin), Antimycobacterials (Rifbutin, Rifampin, Rifapentine) anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals (i.e ketoconazole), or antivirals or antiretroviral (e.g. acyclovir, valacyclovir, Viread®, Atripla®, Emtriva®, or Complera®), St. John's Wort or drugs that may interact with TAF or EVG as specified in the Vitekta and Vemlidy Investigator Brochure, should not be used during the study.
10. Current or anticipated chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetominophen for the duration of the study.
11. Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study
12. Grade 2 or higher laboratory abnormality, per the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
13. Abnormal finding on laboratory or physical examination or a social or medical condition in the volunteer which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Grade 2 or higher treatment-emergent adverse events (TEAEs) | Changes from baseline up to a maximum of 12 days post-dose
  TEAEs are defined as adverse events starting or worsening after administration of the study product; Grade is determined by the DAIDS Grading Table
Number of participants with adverse events | Changes from baseline up to a maximum of 12 days post-dose
  Adverse events for this outcome are those that are product-related urogenital in nature
systemic laboratory assessments | Changes from baseline up to 72 hours post-dose
  Number of participants with abnormal serum chemistry
Systemic Laboratory Assessments | Changes from baseline up to 72 hours post-dose
  Number of participants with abnormal complete blood count
Drug Concentrations of EVG, TFV, and TAF | From dosing to 72 hours post-dose
  Concentrations of EVG, TFV, and TAF in plasma
Drug Concentrations of EVG, TFV, and TAF | From dosing to a maximum of 12 days post-dose
  Concentrations of EVG, TFV, and TAF in CV fluid
Drug Concentrations of EVG, TFV, TFV-DP, and TAF | From dosing to 72 hours post-dose
  Concentrations of EVG, TFV, TFV-DP, TAF in CV tissue

SECONDARY OUTCOMES:
Percent (%) inhibition of HIV in vaginal cell assay (Anti-HIV activity) | Changes from baseline to 24 hours post-dose
  Anti-HIV activity in CV fluid
Percent (%) inhibition of HSV in vaginal cell assay (Anti-HSV activity) | Changes from baseline to 24 hours post-dose
  Anti-HSV activity in CV fluid
Number of participant tissue samples demonstrating HIV-1 infectivity | Changes from baseline to 4 hours post-dose
  p24 antigen production in CV tissue infected with HIV-1 ex vivo
Disintegration of insert | At 4 or 24 hours post-dose (per randomized time point)
  Percent (%) disintegration at the first evaluation after dosing
Acceptability of insert: questionnaire | At baseline and at 48 or 72 hours post-dose (per randomized time point)
  Responses to key questions on acceptability questionnaire (including prior experience with vaginal product use, initial and post-use impressions of insert, dissolution time, discharge amounts, and feelings about real-world use if insert was available for use

OTHER OUTCOMES:
HSV infectivity | Changes from baseline to 24 hours post-dose
  HSV DNA fold change after ex vivo infection of CV tissue with HSV

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — CONRAD
Locations (1):
- Clinical Research Center at Eastern Virginia Medical School (NOT RECRUITING ADDITIONAL SITES), Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurman AR, Ouattara LA, Yousefieh N, Anderson PL, Bushman LR, Fang X, Hanif H, Clark M, Singh O, Doncel GF. A phase I study to assess safety, pharmacokinetics, and pharmacodynamics of a vaginal insert containing tenofovir alafenamide and elvitegravir. Front Cell Infect Microbiol. 2023 Apr 19;13:1130101. doi: 10.3389/fcimb.2023.1130101. eCollection 2023. PMID 37153145